CLINICAL TRIAL: NCT02717091
Title: Phase II Study of Neoadjuvant FOLFIRINOX or Nab-paclitaxel With Gemcitabine for Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant FOLFIRINOX or Nab-paclitaxel With Gemcitabine for Borderline Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, Junpei Yamaguchi, Surgical Oncology, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUDC1508
Record Dates: First submitted 2016-02-11; First posted 2016-03-23 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Borderline Resectable Pancreatic Cancer
MeSH Terms: interventions — folfirinox; Gemcitabine; 130-nm albumin-bound paclitaxel

ARMS (2):
- FOLFIRINOX (Experimental): 4 course of FILFIRINOX before surgery
  Interventions: Drug: FOLFIRINOX
- GEM + nab-PTX (Experimental): 2 course of GEM + nab-PTX before surgery
  Interventions: Drug: gemcitabine + nab-paclitaxel

INTERVENTIONS:
Drug: FOLFIRINOX
  Arms: FOLFIRINOX
Drug: gemcitabine + nab-paclitaxel
  Arms: GEM + nab-PTX

SUMMARY:
The aim of this study is to clarify the efficacy and safety of neoadjuvant FOLFIRINOX and nab-paclitaxel + gemcitabine for borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Borderline resectable pancreatic cancer (based on NCCN guideline version 2.2015)
2. first treatment for pancreatic cancer
3. performance status 0 or 1
4. adequate one marrow function
5. adequate renal function
6. obtained informed consent

Exclusion Criteria:

1. other active concomitant malignancies
2. other severe medical conditions; contraindication of FOLFIRINOX, paclitaxel and gemcitabine
3. pregnant women
4. no informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-06 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3 months
  surgery is supposed to be performed 3 months after the initiation of chemotherapy

SECONDARY OUTCOMES:
completion rate of chemotherapy | 3 months
  chemotherapy is supposed to take 3 months
relative dose intensity | 3 months
  chemotherapy is supposed to take 3 months
adverse event | 3 months
  chemotherapy is supposed to take 3 months
tumor response | 3 months
  tumor response to chemotherapy will be assessed based on Response Evaluation Criteria In Solid Tumor (RECIST). CR: Complete Response, PR: Partial Response, PD: Progression, SD: Stable Disease, NE: Not Evaluable
disease free survival | 3 years after the surgery
overall survival | 3 years after the surgery
surgical complication | 1 month after the surgery
quality of the tumor | 3 months
  Chemotherapy is supposed to take 3 months. After the completion of chemotherapy, the quality of the tumor will be assessed by imaging findings, such as CT number and Standardized uptake value.